CLINICAL TRIAL: NCT00470054
Title: A Phase II Study of Dasatinib (NSC #732517) in Patients With Chemo-Sensitive Relapsed Small Cell Lung Cancer
Brief Title: Dasatinib in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00467; NCI-2009-00467 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000543528; CALGB 30602 (Other: Cancer and Leukemia Group B); CALGB-30602 (Other: CTEP); P30CA014236 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Limited Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Dasatinib

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive oral dasatinib twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Given PO
  Other Names: BMS-354825; Sprycel

SUMMARY:
This phase II trial is studying how well dasatinib works in treating patients with relapse small cell lung cancer. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE I. Determine the efficacy of dasatinib in patients with relapsed small cell lung cancer.

SECONDARY OBJECTIVE II. Determine the objective response rate (complete and partial response) in patients treated with this drug.

III. Determine the overall survival of patients treated with this drug. IV. Determine the toxicity of this drug in these patients.

OUTLINE:

Patients receive oral dasatinib twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at least every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC) (limited or extensive stage disease)
* Progressive or recurrent disease after an initial response to first-line treatment with a platinum-based chemotherapy with or without concurrent definitive radiotherapy to the chest (chemotherapy must have been completed at least 90 days prior to documentation of relapse)
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Lesions that are not considered measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural or pericardial effusion
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Tumor lesions situated in a previously irradiated area, unless progression after radiotherapy is documented in these lesions
* No known brain metastases (previously treated brain metastases allowed provided they are neurologically stable for >= 4 weeks)
* ECOG performance status 0-1
* Platelet count >= 100,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Creatinine =< 1.5 times ULN OR creatinine clearance >= 60 mL/min
* AST =< 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* No significant cardiac disease, including any of the following:

  * New York Heart Association class III-IV heart disease
  * Myocardial infarction or ventricular tachyarrhythmia within the past 6 months
  * Prolonged QTc > 480 msec (Fridericia correction)
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* No more than 1 prior chemotherapy regimen
* No prior dasatinib or compounds of similar chemical composition or similar biologic therapeutic activity including, but not limited to, any inhibitors of SRC, BCR-ABL, c-KIT, EPHA2, or PDGFRB kinases
* At least 2 weeks since prior definitive or palliative radiotherapy (prior radiotherapy allowed in the context of combined modality treatment with curative intent for limited stage disease; prophylactic cranial radiotherapy; or palliative radiotherapy initially or at relapse)
* At least 2 weeks since prior surgery and recovered
* At least 1 week since prior and no concurrent agents with proarrhythmic potential
* At least 1 week since prior and no concurrent CYP3A4 inhibitors or inducers
* At least 1 week since prior and no concurrent grapefruit concentrate
* No concurrent palliative radiotherapy
* No concurrent hormones or other chemotherapeutic agents, except steroids for adrenal failure, hormones for noncancer-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent chemotherapeutic or investigational agents
* Fertile patients must use effective contraception during and for >= 6 weeks after completion of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonius Miller, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2007 and December 2008, 45 participants were recruited.
Pre-assignment Details: One(1) participant cancelled before receiving any protocol related therapy and 1 participant was deemed ineligible. All participants receiving treatment were analyzed for adverse events and only eligible (43) participants were analyzed for al other endpoints.
Groups:
- Dasatinib: Pts receive oral dasatinib 70 mg twice daily
Period: Overall Study
Arm/Group | Dasatinib
Started | 44
Completed | 43
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Only eligible participants (those who met the criteria for inclusion) were evaluated for baseline characteristics.
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 64 [35 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 43
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 12
    1 - Ambulatory, restricted strenuous activity | 31

OUTCOME MEASURES:

1. Primary Outcome: 6 Week Progression Free Survival
Description: Percentage of patients who were alive and progression free at 6-weeks. The 6-week progression free survival was estimated using the Kaplan Meier method.
  Progressive Disease was defined by the Response Evaluation Criteria In Solid Tumors (RECIST) criteria as 20% increase in sum of longest diameter of target lesions.
Time Frame: 6 weeks
Population: All eligible participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
percentage of participants | 43 [30 to 61]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from registration until disease progression or death, whichever occurs first. The median PFS with 95% CI was estimated using the Kaplan-Meier method.
  Progression is defined as in the primary outcome measure.
Time Frame: Time from registration to progression (up to 3 years)
Population: All eligible participants were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
weeks | 5.9 [5.7 to 6.6]

3. Secondary Outcome: Response to Therapy
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Assessed every 2 cycles (up to 3 years)
Population: All eligible participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 7
  Progression | 28
  Inadequately assessed | 8

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death (up to 3 years)
Population: All eligible participants were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
weeks | 17 [14.6 to 29.7]

5. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 was used to evaluate toxicity.
  Grade 1: mild; Grade 2: moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: Assessed during treatment
Population: All 44 participants who received treatment were analyzed (including ineligible participants).
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 44
participants | 12

ADVERSE EVENTS:
Description: All 44 participants who received treatment were analyzed (including ineligible participants).
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 14/44
Other Adverse Events (participants affected / at risk) | 39/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=44)
Hemoglobin (Blood and lymphatic system disorders) | 12 (16)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Death not associated with CTCAE term (General disorders) | 2 (2)
Edema: limb (General disorders) | 4 (4)
Fatigue (General disorders) | 12 (15)
Fever (General disorders) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol serum-high (hypercholesteremia) (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (1)
Lymphopenia (Investigations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 5 (7)
Prolonged QTc interval (Investigations) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4)
Magnesium serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=44)
Hemoglobin (Blood and lymphatic system disorders) | 24 (45)
Lymphatics - Other (Blood and lymphatic system disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 11 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (8)
Death NOS (General disorders) | 1 (1)
Death not associated with CTCAE term (General disorders) | 5 (8)
Edema: limb (General disorders) | 4 (5)
Edema:head and neck (General disorders) | 3 (4)
Fatigue (General disorders) | 34 (62)
Fever (General disorders) | 2 (2)
Syndromes - Other (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (2)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 6 (13)
Prolonged QTc interval (Investigations) | 1 (3)
Weight loss (Investigations) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (15)
Insomnia (Psychiatric disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less